CLINICAL TRIAL: NCT01531504
Title: Evaluation of Safety and Effectiveness of ViKY Device for Uterine Positioning
Brief Title: New Use of the ViKY Device for Uterus Positioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EndoControl (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ViKY UP IDE
Record Dates: First submitted 2012-01-31; First posted 2012-02-13 (Estimated); Last update posted 2012-12-28 (Estimated); Status verified 2012-12

CONDITIONS: Surgical Procedure, Unspecified
Keywords: hysterectomies; uterine manipulator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hysterectomy (Other): candidate for a conventional laparoscopic-assisted
  Interventions: Device: ViKY UP

INTERVENTIONS:
Device: ViKY UP — laparoscopic-assisted hysterectomy procedure

SUMMARY:
Evaluation of Safety and Efficacy of ViKY Device for Uterus Positioning on 2 US sites

DETAILED DESCRIPTION:
The ViKY device "Vision Control for endoscopy" was initially a compact motorized endoscope holder for laparoscopic surgery. It holds the endoscope and is controlled by either a foot pedal or voice activation. It received FDA approval in December 2008 and since that time has been used to facilitate laparoscopic surgery in multiple specialties.

EndoControl now considers using the technology for uterus manipulation in laparoscopic-assisted hysterectomies. Most gynecologic surgeries require displacement of the uterus out of the anatomic location to optimize the surgery. During an abdominal hysterectomy clamps are placed on the uterine cornua allowing easy manipulation of the uterus. The development of laparoscopic surgery required new techniques to manipulate the uterus. Typically a uterine manipulator is placed vaginally and controlled by the surgeon or the surgical assistant during the procedure.

In conventional operations, the constant physical force decreases the surgical team's efficacy and increases fatigue levels. The use of the ViKY device to control the position of the uterus facilitates surgery by enabling the surgeon to maintain a constant "locked" position or by allowing the surgeon to remotely move the uterus at any point of the surgery. The ViKY device also eliminates the need for an extra surgical assistant during laparoscopic-assisted hysterectomies.

The aim of this study is to collect data to demonstrate safety and effectiveness of the use of the ViKY device for uterine manipulation during conventional laparoscopic-assisted hysterectomies or computer-controlled laparoscopic hysterectomies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Candidate for conventional laparoscopic-assisted hysterectomies procedures
* patient has a cervix and a uterus

Exclusion criteria

* Difficulty understanding the English language
* Anatomy that precludes the use of a uterine manipulator
* Current inclusion in another research study

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-12; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Effectiveness | 4 months
  Number of cases with adequate visualization of pelvic anatomy during endoscopy.
Adverse Events | 4 months
  Number of perforations during intervention. Number of complications associated with the use of uterine manipulator

SECONDARY OUTCOMES:
surgery characterization | 4 months
  Duration of time of each procedure, duration of time to set up Viky UP device

CONTACTS AND LOCATIONS:
Overall Officials: Arnold ADVINCULA, MD, Principal Investigator — Floridal Hospital; Kevin STEPP, MD, Principal Investigator — Carolinas Medical Center
Locations (2):
- United States (2):
  - Florida Hospital, Orlando, Florida
  - Carolinas Medical Center, Charlotte, North Carolina